CLINICAL TRIAL: NCT05556083
Title: Efficacy of Adding Sildenafil to Dapoxetine in Treatment of Dapoxetine Non-responding Mono-symptomatic Premature Ejaculation (PE)
Brief Title: Sildenafil Added Effect in Dapoxetine Non-responding Mono-symptomatic Premature Ejaculation (PE)
Acronym: PE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Almetwally Algammal,MD, Clinical professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61158m1
Record Dates: First submitted 2022-09-10; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Premature Ejaculation
Keywords: Premature ejaculation; Sildinafile; Dapoxitine
MeSH Terms: conditions — Premature Ejaculation | interventions — Sildenafil Citrate; Tablets

STUDY DESIGN:
Intervention Model Description: Single blind placebo randomized controlled trial
Who Masked: Participant
Masking Description: participants of both groups will have no knowlage regarding the added medication they will recieve either sildinafile or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sofenacine recievers group A (Active Comparator): Group (A) will receive sildenafil 50mg tablet form as additive therapy to dapoxetine 30 mg tablet form on demand for 8 weeks.
  Interventions: Drug: Sildenafil 50 mg Oral Tablet and Dapoxitine 3mg Oral tablet
- palcebo recievers group B (Placebo Comparator): Group (B) will continue on dapoxetine 30mg tablet form with placebo tablet form of the same shap and colour of sildinafile on demand for 8 weeks.
  Interventions: Drug: Placebo oral tablet and Dapoxitine 3mg Oral tablet

INTERVENTIONS:
Drug: Sildenafil 50 mg Oral Tablet and Dapoxitine 3mg Oral tablet — Single blind placebo randomized controlled trial
  Other Names: viagra; prigily
  Arms: sofenacine recievers group A
Drug: Placebo oral tablet and Dapoxitine 3mg Oral tablet — Single blind placebo randomized controlled trial
  Arms: palcebo recievers group B

SUMMARY:
Study Design: Single Blind Placebo Controlled Randomized Trial, aiming to assess the efficacy and safety of adding sildinafile 50 mg to dapoxitine 30 mg in dapoxitine non responding premature ejaculation.

DETAILED DESCRIPTION:
Study Design: Single Blind, Placebo Controlled Randomized Trial.

Study Setting: Urology outpatient clinics at Al-Hussein and Sayed Galal Hospitals; Al-Azhar University; Cairo; Egypt.

Timeline: 12 months [8 months for data collection; 2 months for thesis writing and 2 months for publication].

Study Population:

* The study participants will be males suffering from primary or acquired mono-symptomatic premature ejaculation (PE) that did not respond to 2 months of dapoxetine monotherapy.
* participants will considered to have PE if they fulfilled the criteria of the International Society for Sexual Medicine that defines PE as a male sexual dysfunction characterized by (i) ejaculation which always or nearly always occurs prior to or within 1 min of vaginal penetration, either present from the first sexual experience or following a new bothersome change in ejaculatory latency. (ii) Negative personal consequences, such as distress, bother, frustration and/or the avoidance of sexual intimacy(Gillman & Gillman, 2019).
* Other patient inclusion criteria will be: age ≥20 years old, married and in a stable regular sexual relationship for at least 3 months before the study.

Exclusion criteria:

* Men with associated erectile dysfunction (ED).
* Men with associated chronic prostatitis.
* Diabetes Mellitus (DM).
* Advanced renal or hepatic diseases.
* Neurological diseases and C.N.S. medications.
* Contraindication to sildenafil as Nitric Oxide dependent ischemic heart disease patients or drug allergy.

Study Sample:

- All available cases with complete medical record and accepted follow-up with us will be included.

Study Procedures and Data Collection:

* Single blind placebo randomized controlled trial will be conducted on 200 male participants with PE divided into two groups 100 participant in each.
* The participants will be selected from those seeking medical advice at the outpatient clinics of Al-Hussein and Sayed Galal Hospitals; Al-Azhar University; Cairo; Egypt starting from October 2022.
* An informed consent will be obtained by each participant after full explanation for the nature of the research.
* The medical records of all adult males suffering from mono-symptomatic premature ejaculation who were treated with on demand dapoxetine for 2 months with no improvement and agree to participate in the study will be reviewed for,

  1. Demographic and clinical data as, age, comorbidities, occupation, parity, body mass index.
  2. Detailed medical and sexual history.
  3. All patients will be evaluated by the International Index of Erectile Function 5 (IIEF5) item questionnaires to exclude those with erectile dysfunction (score ≥22) and premature ejaculation diagnostic tool (PEDT).
  4. Physical examination including local abdominal and genital examination.
  5. Urine analysis with culture and sensitivity.
  6. Abdominopelvic ultrasonography.
  7. If needed Penile duplex US and Or Nocturnal Penile Tumescence and Rigidity (NPTR)will be performed to exclude organic ED.

     Participants of our study will be enrolled into two groups (A and B). participants enrollment will be done by simple randomization method through which none of participants know in which group he will be. Group (A) will receive sildenafil 50mg as additive therapy to dapoxetine 30 mg for 8 weeks. Group (B) will continue on dapoxetine 30mg with placebo for the same period as group (A).

     All patients will be instructed to do sexual intercourse 2-3 times a week.
* All patients were evaluated before and after the treatment by Premature Ejaculation Diagnostic Tool (PEDT) and IIEF-5, using the validated Arabic version of both questionnaires, Questionnaire will be fulfilled by face to face interview method.

Protection of Participants:

1. The research will be explained in detail to the participants before inclusion in the study.
2. Participants will sign an informed written consent before enrollment.
3. Extreme care will be taken during the research related procedures.
4. It will be made clear that the subject has the full right to withdraw from the study at any time.
5. Informed consent and all study material will be kept in separate lockers; not accessed except by study investigators.

ELIGIBILITY:
Inclusion Criteria:

* Male patients, age ≥20 years old, married and/or in a stable regular sexual relationship for at least 3 months before the study.

Exclusion Criteria:

* - Men with associated erectile dysfunction (ED).
* Men with associated chronic prostatitis.
* Diabetes Mellitus (DM).
* Advanced renal or hepatic diseases.
* Neurological diseases and C.N.S. medications.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-09-29 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
intravaginal latency time changes IVLT | Eight weaks for each participant of both groups
  Using PEDT premature ejaculation diagnostic tool (PEDT)
overall partner satisfaction | Eight weaks for each participants of both groups
  using Sexual Satisfaction Index (SSI).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Algammal, MD., Principal Investigator — urologist